CLINICAL TRIAL: NCT04056117
Title: Safety and Immunogenicity of a Shigella-Tetravalent Bioconjugate Vaccine: A Phase 1/2 Randomized Controlled and Age Descending Study Including Dose Finding in 9 Month Old Infants
Brief Title: A Study to Determine If a New Shigella Vaccine is Safe, Induces Immunity and The Best Dose Among Kenyan Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LimmaTech Biologics AG (Industry)
Collaborators: Kenya Medical Research Institute (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S4V01
Record Dates: First submitted 2019-07-26; First posted 2019-08-14 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Shigellosis
MeSH Terms: conditions — Dysentery, Bacillary | interventions — MenACWY; Tetanus Toxoid

STUDY DESIGN:
Intervention Model Description: This phase 1/2 trial is a multicentre, randomized, controlled, double blind, with two steps; a step 1 with a safety cohort and a step 2 with a dose-finding cohort. Safety of the vaccine will be evaluated first in adults and subsequently in children and infants through an age-descending and dose escalation approach (safety cohort, step 1). Following confirmation of vaccine safety, further cohorts of infants (dose-finding cohort) will be enrolled to evaluate immunogenicity of the vaccine at different doses and expand safety data (step 2). Vaccination in Step 1 will be staggered with adults being the first to be vaccinated and infants last. In step 2 infants will be vaccinated concurrently, with each group randomised to receive 1 of 4 different vaccine doses. A control vaccine will be used, and participants will be randomized at a ratio of 3:1 in adults, 2:1 in children, 2:1 in infants in step 1 and 8:1 in infants in step 2, to receive the candidate vaccine versus the control vaccine.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (19):
- NA (Non-adjuvanted) - very low dose - infants (Experimental): Infants receive 3 very low doses of the non-adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- A (adjuvanted) - very low dose - infants (Experimental): Infants receive 3 very low doses of the adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- NA (Non-adjuvanted) - low dose -infants (Experimental): Infants receive 3 low doses of the non-adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- A (adjuvanted) - low dose - infants (Experimental): Infants receive 3 low doses of the adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- NA (non-adjuvanted) - medium dose - infants (Experimental): Infants receive 3 medium doses of the non-adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- A (adjuvanted) - medium dose - infants (Experimental): Infants receive 3 medium doses of the adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- NA (non-adjuvanted) - medium dose - children (Experimental): Children receive 3 medium doses of the non-adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- A (adjuvanted) - medium dose - children (Experimental): Children receive 3 medium doses of the adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- NA (non-adjuvanted) - medium dose-adults (Experimental): Adults receive 2 medium doses of the non-adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- A (adjuvanted) - medium dose - adults (Experimental): Adults receive 2 medium doses of the adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- NA (non-adjuvanted) - high dose - infants (Experimental): Infants receive 3 high doses of the non-adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- A (adjuvanted) - high dose - infants (Experimental): Infants receive 3 high doses of the adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- NA (non-adjuvanted) - high dose - children (Experimental): Chilldren receive 3 high doses of the non-adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- A (adjuvanted) - high dose - children (Experimental): Chilldren receive 3 high doses of the adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- NA (non-adjuvanted) - high dose - adults (Experimental): Adults receive 2 high doses of the non-adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- A (adjuvanted) - high dose - adults (Experimental): Adults receive 2 high doses of the adjuvanted investigational product
  Interventions: Biological: Shigella 4V
- MenACWY-Placebo (Experimental): Adults receive one administration of MenACWY followed by one placebo administration
  Interventions: Biological: MenACWY; Biological: Placebo
- Rabies (Other): Children receive three administrations of Rabies
  Interventions: Biological: Rabies
- MenACWY-DTaP (Other): Infants receive two administrations of MenACWY followed by DTaP administration
  Interventions: Biological: MenACWY; Biological: Diphtheria, Tetanus and Pertussis (DTaP)

INTERVENTIONS:
Biological: Shigella 4V — Non-adjuvanted and adjuvanted Shigella 4V administrated at 4 different doses: very low, low, medium and high.
  Arms: A (adjuvanted) - high dose - adults; A (adjuvanted) - high dose - children; A (adjuvanted) - high dose - infants; A (adjuvanted) - low dose - infants; A (adjuvanted) - medium dose - adults; A (adjuvanted) - medium dose - children; A (adjuvanted) - medium dose - infants; A (adjuvanted) - very low dose - infants; NA (Non-adjuvanted) - low dose -infants; NA (Non-adjuvanted) - very low dose - infants; NA (non-adjuvanted) - high dose - adults; NA (non-adjuvanted) - high dose - children; NA (non-adjuvanted) - high dose - infants; NA (non-adjuvanted) - medium dose - children; NA (non-adjuvanted) - medium dose - infants; NA (non-adjuvanted) - medium dose-adults
Biological: MenACWY — Control vaccine administrated to adults and infants
  Arms: MenACWY-DTaP; MenACWY-Placebo
Biological: Rabies — Control vaccine administrated to children
  Arms: Rabies
Biological: Diphtheria, Tetanus and Pertussis (DTaP) — Control vaccine administrated to infants
  Arms: MenACWY-DTaP
Biological: Placebo — Control administrated to adults
  Arms: MenACWY-Placebo

SUMMARY:
In this study, the tetravalent bioconjugate candidate vaccine Shigella4V will be tested to obtain first-in-human data on its safety and immunogenicity in infants and to identify the preferred dose of Shigella4V in 9 month old infants.

DETAILED DESCRIPTION:
Shigella4V is a tetravalent bioconjugate vaccine including O antigen-polysaccharides of the most predominant Shigella serotypes.

The study will be conducted in two steps. In Step1: safety and reactogenicity of the vaccine will be evaluated first in adults and subsequently in children and infants through an age-descending and dose escalation approach. In Step 2: in order to further evaluate safety and to identify the optimum immunogenic dose, infants will be randomised to receive 1 of 4 different vaccine doses or control vaccine.

Adults will receive a 2 dose schedule, children and infants will receive a 3 dose schedule. For each vaccine dose, formulation with and without Aluminium adjuvant will be tested.

ELIGIBILITY:
Inclusion Criteria:

All ages

* Healthy by medical history, laboratory findings and physical examination before entering into the study (Participants with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator)
* Seronegative for HIV, hepatitis B and C (as per screening laboratory tests)
* Resident in the study area village during the whole trial period (Kilifi -Kilifi Health and Demographic Surveillance System (Described in more detail in the SSA); (Kericho-a 75km radius from the Kericho Clinical Research Centre).
* Previously completed routine primary vaccinations (6,10 and 14 weeks or thereabouts) to the best knowledge of the participant/parent/guardian.
* Signed/thumb written informed consent, in accordance with local practice, provided by adult volunteers (participants 18 years of age and older), parents or legal representatives for children and infants participants as applicable, who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* Demonstrated comprehension of the protocol procedures by passing score of 90% or better on a written/verbal comprehension test.

Adults

* Female and male participants between, and including 18-50 years at the time of first vaccination
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause. Female volunteers of childbearing potential may be enrolled in the study if the participant: has a negative urine pregnancy test at the day of screening and vaccinations, respectively, and

  * agree to use effective contraception for 30 days prior to vaccination and
  * agree to continue contraception at least for 2 months after completion of vaccination series.

Children and Infants

* Female and male aged 9 months (+/- 1 month) old (infants) or between, and including, 2-5 years of age (children) at the time of the first vaccination
* Born full-term (i.e. after a gestation period of 37 to less than 42 completed weeks)

Exclusion Criteria:

All ages

* Any clinically significant deviation from the normal range in biochemistry or haematological blood tests.
* Suspected or known hypersensitivity (including allergy) to any of the vaccine components or to previous vaccine, or to medicinal products or medical equipment whose use is foreseen in this study
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws
* Any confirmed or suspected immunosuppressive or immune-deficient condition.
* Systemic administration of corticosteroids (PO/IV/IM): prednisone ≥20 mg/day, or equivalent for more than 14 consecutive days from birth (for infants) / within 90 days prior to informed consent. Inhaled except for doses > 800 mg/day and topical steroids are allowed.
* Administration of antineoplastic or radiotherapy from birth / within 90 days prior to informed consent. Participants may be on chronic or as needed medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition
* Known exposure to Shigella during lifetime of the subject
* Concurrently participating in another clinical study, or participation in the preceding month, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device)
* Acute disease and /or fever at the time of enrolment Note: enrolment may be postponed/delayed until such transient circumstances have terminated
* History of any malignancy of lymphoproliferative disorder
* Known to be part of study personnel or being a close family member to the personnel conducting this study.
* Previous history of significant persistent neutropenia, or drug related Neutropenia
* Adults with clinical wasting; children with weight-for-age Z score less than -3SD.
* History of any chronic or progressive disease (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease) that according to judgment of the investigator could interfere with the study outcomes or pose a threat to the participant's health
* History of surgical splenectomy or Sickle cell disease (SCD test performed at KEMRI-CGMRC only).
* Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine
* Any medical, social condition, or occupational reason that, in the judgment of the investigator, is a contraindication to protocol participation or impairs the volunteer's/parent's/guardian's ability to give informed consent, increases the risk to the potential participant because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data .

Adults

* Women who are breastfeeding
* History of chronic alcohol consumption and/or drug abuse. Chronic alcohol consumption is defined as: a prolonged period of frequent, heavy alcohol use; the inability to control drinking once it has begun; physical dependence manifested by withdrawal symptoms when the individual stops using alcohol; tolerance, or the need to use more and more alcohol to achieve the same effects; a variety of social and/or legal problems arising from alcohol use.

Ages: 8 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 596 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Safety - Solicited Local and Systemic Adverse Events (AEs) | during 7 days following each vaccination
  Safety and tolerability of the candidate vaccine Shigella4V as determined by occurrence, severity and relationship of solicited AEs
Safety - Unsolicited Adverse Events (AEs) | during 28 days following each vaccination
  Safety and tolerability of the candidate vaccine Shigella4V as determined by occurrence, severity and relationship of unsolicited AEs
Safety - Serious Adverse Events (SAEs) | throughout the study duration, up to 15 months
  Safety and tolerability of the candidate vaccine Shigella4V as determined by occurrence, severity and relationship of SAEs
Immunology - change in serum immunoglobulin G (IgG) | throughout the study, up to 15 months
  Serum IgG responses and fold-increases between post- and pre-vaccination samples from infants of step 2, as determined by enzyme-linked immunosorbent assay (ELISA) against lipopolysaccharide (LPS) corresponding to the 4 Shigella serotypes included in the Shigella4V bioconjugate.

SECONDARY OUTCOMES:
Safety - clinically significant changes in cell blood count (CBC) with differentials | throughout the study, up to 15 months
  Assess the safety of the candidate vaccine Shigella4V by measuring clinical significant changes in haematological safety parameters
Safety - clinically significant changes in creatinine level | throughout the study, up to 15 months
  Assess the safety of the candidate vaccine Shigella4V by measuring clinical significant changes in biochemical safety parameters
Safety - clinically significant changes in alanine aminotransferase (ALT) level | throughout the study, up to 15 months
  Assess the safety of the candidate vaccine Shigella4V by measuring clinical significant changes in biochemical safety parameters
Safety - clinically significant changes in aspartate aminotransferase (AST) level | throughout the study, up to 15 months
  Assess the safety of the candidate vaccine Shigella4V by measuring clinical significant changes in biochemical safety parameters
Immunogenicity - change is serum IgG | throughout the study, up to 15 months
  Serum IgG responses and fold-increases between post- and pre-vaccination samples from all participants of step 1, as determined by ELISA against LPS corresponding to the 4 Shigella serotypes included in the Shigella4V bioconjugate.
Immunogenicity - change in anti-Shigella LPS antibody titre | throughout the study, up to 15 months
  Percentage of participants (from step 1 and 2) achieving at least a four-fold rise in anti-Shigella LPS antibody titre after each injection compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mainga Hamaluba, MD, Principal Investigator — KEMRI/Welcome Trust Research Programme,Kilifi, Kenya; Josphat Kosgei, MD, Principal Investigator — Medical Research Institute, Kericho, Kenya
Locations (2):
- Kenya (2):
  - Kenya Medical Research Institute (KEMRI)/ United States Army Medical Research Directorate- Kenya (USAMRD-K), Kericho
  - KEMRI-Centre Geographic Medical Research-COAST (KEMRI-CGMRC), Kilifi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2015 LRI Collaborators. Estimates of the global, regional, and national morbidity, mortality, and aetiologies of lower respiratory tract infections in 195 countries: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Infect Dis. 2017 Nov;17(11):1133-1161. doi: 10.1016/S1473-3099(17)30396-1. Epub 2017 Aug 23. PMID 28843578
- [Background] Livio S, Strockbine NA, Panchalingam S, Tennant SM, Barry EM, Marohn ME, Antonio M, Hossain A, Mandomando I, Ochieng JB, Oundo JO, Qureshi S, Ramamurthy T, Tamboura B, Adegbola RA, Hossain MJ, Saha D, Sen S, Faruque AS, Alonso PL, Breiman RF, Zaidi AK, Sur D, Sow SO, Berkeley LY, O'Reilly CE, Mintz ED, Biswas K, Cohen D, Farag TH, Nasrin D, Wu Y, Blackwelder WC, Kotloff KL, Nataro JP, Levine MM. Shigella isolates from the global enteric multicenter study inform vaccine development. Clin Infect Dis. 2014 Oct;59(7):933-41. doi: 10.1093/cid/ciu468. Epub 2014 Jun 23. PMID 24958238
- [Background] Mani S, Wierzba T, Walker RI. Status of vaccine research and development for Shigella. Vaccine. 2016 Jun 3;34(26):2887-2894. doi: 10.1016/j.vaccine.2016.02.075. Epub 2016 Mar 12. PMID 26979135
- [Background] Ashkenazi S, Cohen D. An update on vaccines against Shigella. Ther Adv Vaccines. 2013 Sep;1(3):113-23. doi: 10.1177/2051013613500428. PMID 24757519
- [Background] Kotloff KL, Nataro JP, Blackwelder WC, Nasrin D, Farag TH, Panchalingam S, Wu Y, Sow SO, Sur D, Breiman RF, Faruque AS, Zaidi AK, Saha D, Alonso PL, Tamboura B, Sanogo D, Onwuchekwa U, Manna B, Ramamurthy T, Kanungo S, Ochieng JB, Omore R, Oundo JO, Hossain A, Das SK, Ahmed S, Qureshi S, Quadri F, Adegbola RA, Antonio M, Hossain MJ, Akinsola A, Mandomando I, Nhampossa T, Acacio S, Biswas K, O'Reilly CE, Mintz ED, Berkeley LY, Muhsen K, Sommerfelt H, Robins-Browne RM, Levine MM. Burden and aetiology of diarrhoeal disease in infants and young children in developing countries (the Global Enteric Multicenter Study, GEMS): a prospective, case-control study. Lancet. 2013 Jul 20;382(9888):209-22. doi: 10.1016/S0140-6736(13)60844-2. Epub 2013 May 14. PMID 23680352
- [Background] Anderson M, Sansonetti PJ, Marteyn BS. Shigella Diversity and Changing Landscape: Insights for the Twenty-First Century. Front Cell Infect Microbiol. 2016 Apr 19;6:45. doi: 10.3389/fcimb.2016.00045. eCollection 2016. PMID 27148494
- [Background] Kotloff KL, Platts-Mills JA, Nasrin D, Roose A, Blackwelder WC, Levine MM. Global burden of diarrheal diseases among children in developing countries: Incidence, etiology, and insights from new molecular diagnostic techniques. Vaccine. 2017 Dec 14;35(49 Pt A):6783-6789. doi: 10.1016/j.vaccine.2017.07.036. Epub 2017 Jul 29. PMID 28765005
- [Background] Juergens C, de Villiers PJ, Moodley K, Jayawardene D, Jansen KU, Scott DA, Emini EA, Gruber WC, Schmoele-Thoma B. Safety and immunogenicity of 13-valent pneumococcal conjugate vaccine formulations with and without aluminum phosphate and comparison of the formulation of choice with 23-valent pneumococcal polysaccharide vaccine in elderly adults: a randomized open-label trial. Hum Vaccin Immunother. 2014;10(5):1343-53. doi: 10.4161/hv.27998. Epub 2014 Feb 27. PMID 24576885
- [Background] Bryant K, McVernon J, Marchant C, Nolan T, Marshall G, Richmond P, Marshall H, Nissen M, Lambert S, Aris E, Mesaros N, Miller J. Immunogenicity and safety of measles-mumps-rubella and varicella vaccines coadministered with a fourth dose of Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine in toddlers: a pooled analysis of randomized trials. Hum Vaccin Immunother. 2012 Aug;8(8):1036-41. doi: 10.4161/hv.20357. Epub 2012 Aug 1. PMID 22617844
- [Background] Miller E, Andrews N, Waight P, Findlow H, Ashton L, England A, Stanford E, Matheson M, Southern J, Sheasby E, Goldblatt D, Borrow R. Safety and immunogenicity of coadministering a combined meningococcal serogroup C and Haemophilus influenzae type b conjugate vaccine with 7-valent pneumococcal conjugate vaccine and measles, mumps, and rubella vaccine at 12 months of age. Clin Vaccine Immunol. 2011 Mar;18(3):367-72. doi: 10.1128/CVI.00516-10. Epub 2010 Dec 29. PMID 21191076
- [Background] Taylor DN, Trofa AC, Sadoff J, Chu C, Bryla D, Shiloach J, Cohen D, Ashkenazi S, Lerman Y, Egan W, et al. Synthesis, characterization, and clinical evaluation of conjugate vaccines composed of the O-specific polysaccharides of Shigella dysenteriae type 1, Shigella flexneri type 2a, and Shigella sonnei (Plesiomonas shigelloides) bound to bacterial toxoids. Infect Immun. 1993 Sep;61(9):3678-87. doi: 10.1128/iai.61.9.3678-3687.1993. PMID 8359890
- [Background] Ashkenazi S, Passwell JH, Harlev E, Miron D, Dagan R, Farzan N, Ramon R, Majadly F, Bryla DA, Karpas AB, Robbins JB, Schneerson R. Safety and immunogenicity of Shigella sonnei and Shigella flexneri 2a O-specific polysaccharide conjugates in children. J Infect Dis. 1999 Jun;179(6):1565-8. doi: 10.1086/314759. PMID 10228084